CLINICAL TRIAL: NCT03476668
Title: Relationship Between Dopaminergic Asymmetric Degeneration and Attentional Resources in Parkinson's Disease.
Acronym: RTsAsMIRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Generale Di Zona Moriggia-Pelascini (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MIRT-RTs-Laterality
Record Dates: First submitted 2018-03-19; First posted 2018-03-26 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Parkinson Disease; Attention Disturbances
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RPD PD patients (Active Comparator): Right-side affected PD patients. Intervention: MIRT
  Interventions: Other: MIRT
- LPD PD patients (Active Comparator): Left-side affected (LPD) PD patients. Intervention: MIRT
  Interventions: Other: MIRT

INTERVENTIONS:
Other: MIRT — 4-week multidisciplinary intensive rehabilitation treatment

SUMMARY:
The researchers aimed to investigate the relationship between the asymmetric dopaminergic degeneration and the attentional resources in a group of patients with Parkinson's disease (PD).

DETAILED DESCRIPTION:
To bypass the impaired habitual motor-behavioural control, Parkinson's disease (PD) patients may exploit the network of goal-directed mode of action. The frontostriatal connections underline this functioning, that is based on attention. Since the cognitive processes are related with dopamine, the asymmetrical degeneration of the dopaminergic system affects differently the right side affected (RPD) and the left side affected (LPD) PD patients.

The aim of the study was to investigate the relationship between the asymmetric dopaminergic degeneration and the attentional resources in a group of patients with PD.

ELIGIBILITY:
Inclusion Criteria:

* Stage 2.5-3 according to the Hoehn and Yahr scale (H&Y);
* Stable pharmacological treatment for the last 6 weeks before the enrolment and during the hospitalization;
* Mini Mental State Examination (MMSE) ≥ 24;
* No evidences of dysexecutive syndrome.

Exclusion Criteria:

* Any focal brain lesion detected in brain imaging studies (CT or MRI) performed in the previous 12 months;
* Drug-induced dyskinesias;
* Disturbing resting and/or action tremor, corresponding to scores 2-4 in the specific items of UPDRS III;
* Behavioral disturbances (evaluated with Neuropsychiatric Inventory);
* Visual and auditory dysfunctions according to the general clinical evaluation and medical history;
* Equivocal report about the side of disease onset or bilateral motor involvement.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
Visual Reaction Times (V RTs) | 4 weeks
  Visual Reaction Times
Auditory Reaction Times (A RTs) | 4 weeks
  Auditory Reaction Times
Multiple Choices RTs (MC RTs) | 4 weeks
  Multiple Choices RTs

SECONDARY OUTCOMES:
Unified Parkinson's Disease Rating Scale (UPDRS) | 4 weeks
  Unified Parkinson's Disease Rating Scale
Timed Up and Go Test (TUG) | 4 weeks
  Timed Up and Go Test

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Frazzitta, MD, Principal Investigator — epartment of Parkinson's disease, Movement Disorders and Brain Injury Rehabilitation, "Moriggia-Pelascini" Hospital - Via Pelascini, 3, 22015, Gravedona ed Uniti, Como, Italy

IPD SHARING:
Plan to Share IPD: No